CLINICAL TRIAL: NCT03111550
Title: Clinical Investigation of the TECNIS Next-Generation Intraocular Lens
Brief Title: Clinical Investigation of the Next-Generation Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDOF-121-NGPC
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: subject/evaluator-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Investigational Lens Device #1 (Other): Investigational Intraocular Lens Device #1: Tecnis Model ZHR00
  Interventions: Device: Investigational Intraocular Lens Device #1: TECNIS Model ZHR00
- Investigational Lens Device #2 (Other): Investigational Intraocular Lens Device #2: Tecnis Model ZQR00
  Interventions: Device: Investigational Intraocular Lens Device #2: TECNIS Model ZQR00
- Control Device (Other): Control TECNIS Symfony® Extended Range of Vision Intraocular Lens: Model ZXR00
  Interventions: Device: TECNIS Symfony® Extended Range of Vision Intraocular Lens: Model ZXR00

INTERVENTIONS:
Device: Investigational Intraocular Lens Device #1: TECNIS Model ZHR00 — Intraocular lens replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #1
Device: Investigational Intraocular Lens Device #2: TECNIS Model ZQR00 — Intraocular lens replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #2
Device: TECNIS Symfony® Extended Range of Vision Intraocular Lens: Model ZXR00 — Intraocular lens replaces the natural lens removed during cataract surgery.
  Arms: Control Device

SUMMARY:
This study is a 6-month, prospective, multicenter, bilateral, randomized clinical investigation of the TECNIS Model ZHR00 and Model ZQR00 IOLs versus the TECNIS Symfony control IOL.

The study was conducted at 12 sites in the U.S.A and treated approximately 240 subjects, equally split between the two test groups and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts
* Potential for postoperative BCDVA of 20/30 Snellen or better
* Corneal astigmatism of 1.00 D or less in both eyes
* Normal corneal topography
* Clear intraocular media other than cataract in each eye
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries

Exclusion Criteria:

* Any clinically-significant pupil abnormalities (non-reactive, fixed pupils, or abnormally-shaped pupils)
* Irregular corneal astigmatism
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study
* Inability to achieve keratometric stability for contact lens wearers
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Subjects with diagnosed degenerative visual disorders
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use of tamsulosin or silodosin
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness
* Known ocular disease or pathology that may affect visual acuity or may require surgical intervention during the course of the study or may be expected to require retinal laser treatment or other surgical intervention during the course of the study
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 45 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devi Priya Janakiraman, OD,FAAO, Study Director — Abbott Medical Optics
Locations (12):
- United States (12):
  - Empire Eye and Laser Center, Bakersfield, California
  - Assil Eye Institute, Beverly Hills, California
  - Jones Eye Care, Sioux City, Iowa
  - Chesapeake Eye Care and Laser, Annapolis, Maryland
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Ophthalmology Consultants LTD, St Louis, Missouri
  - Scott and Christie and Associates,PC, Cranberry Township, Pennsylvania
  - Carolina Cataract and Laser Center, Ladson, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Key-Whitman Eye Center, Dallas, Texas
  - Texas Eye and Laser Center, Hurst, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 242 subjects were enrolled in this study, and 229 subjects were implanted with study IOL in first eye.
Groups:
- Tecnis ZHR00; Tecnis ZQR00: Investigational Lens Device
- Tecnis ZXR00: Control Lens Device
Period: Overall Study
Arm/Group | Tecnis ZHR00 | Tecnis ZQR00 | Tecnis ZXR00
Started | 77 (First eye) | 73 (First eye) | 79 (First eye)
Completed | 73 | 71 | 76
Not Completed | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecnis ZHR00 | Tecnis ZQR00 | Tecnis ZXR00 | Total
Number analyzed (Participants) | 77 | 73 | 79 | 229
Age, Customized [Number; unit: Participants]
  Les than < 60 years | 10 | 11 | 7 | 28
  60-69 years | 37 | 34 | 44 | 115
  70-79 years | 29 | 24 | 27 | 80
  Greater than or equal to >= 80 years | 1 | 4 | 1 | 6
  Not reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 46 | 141
  Male | 29 | 26 | 33 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 76 | 71 | 77 | 224
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (including Indian) | 3 | 2 | 1 | 6
  Black | 2 | 2 | 5 | 9
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0
  Caucasian | 71 | 69 | 73 | 213
  Other race | 1 | 0 | 0 | 1
  Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Distance Corrected Near Visual Acuity (DCNVA) at 40 cm
Description: The primary effectiveness endpoint is mean (LogMAR), photopic, monocular, first-eye, distance corrected near visual acuity (40 cm) at 1 month postoperative
Time Frame: 1 month postoperative
Population: The safety population (SP) of all subjects implanted who have available data will be used for all analysis. For the monocular endpoints, the safety population will consist of first eyes implanted with a study IOL.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Tecnis ZHR00 | Tecnis ZQR00 | Tecnis ZXR00
Number analyzed (Participants) | 76 | 72 | 78
Number analyzed (Eyes) | 76 | 72 | 78
LogMAR | 0.136 (0.120) | 0.141 (0.149) | 0.276 (0.116)

2. Primary Outcome: Rates of Adverse Events vs ISO (International Organization for Standardization) SPE ( Safety and Performance Endpoint) Rates (6-Month Persistent Medical Complications/Adverse Events vs ISO 11979-9 SPE Rates)
Description: Adverse Event rates for the Models ZHR00 and ZQR00 investigational lens first eyes are compared to the ISO (International Organization for Standardization) SPE (Safety and performance Endpoint) rates using a one-sided, exact test based on the binomial distribution.
  ISO (the International Organization for Standardization) is a worldwide federation of national standards bodies (ISO member bodies).
  ISO 11979-7 is a document that specifies the particular requirements for the clinical investigations of intraocular lenses that are implanted in the eye in order to correct aphakia.
  SPE rate: safety and performance endpoint (rate derived from analysis of the data from clinical investigations of IOLs approved in the US).
  Only AE rates that are higher than ISO SPE rate value are required to do statistical comparison. Any AE rate that is below ISO SPE value, statistical testing is not necessary to see if the rate is significantly higher than ISO.
Time Frame: 6 months postoperative
Population: Statistical comparisons to ISO SPE rates are based on first-eye data
Measure: Number; unit: Percent
Arm/Group | Tecnis ZHR00 | Tecnis ZQR00 | Tecnis ZXR00
Number analyzed (Participants) | 73 | 71 | 76
Percent
  Corneal edema | 0.0 | 0.0 | 1.3
  Cystoid macular edema | 0.0 | 0.0 | 0.0
  Iritis | 0.0 | 0.0 | 0.0
  Raised IOP requiring treatment | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Tecnis ZXR00; Test type: Superiority — Compare if study AE rate is significantly higher than ISO SPE rate (0.3% for corneal edema); p = 0.02041, Exact test on binomial distribution

3. Primary Outcome: Rates of Adverse Events vs ISO SPE Rates (6-Month Cumulative Medical Complications/Adverse Events vs ISO 11979-9 SPE Rates)
Description: Adverse Event rates for the Models ZHR00 and ZQR00 investigational lens first eyes are compared to the ISO SPE rates using a one-sided, exact test based on the binomial distribution.
  Only AE rates that are higher than ISO SPE rate value are required to do statistical comparison. Any AE rate that is below ISO SPE value, statistical testing is not necessary to see if the rate is significantly higher than ISO.
Time Frame: 6 months postoperative
Population: Statistical comparisons to ISO SPE rates are based on first-eye data
Measure: Number; unit: Percent
Arm/Group | Tecnis ZHR00 | Tecnis ZQR00 | Tecnis ZXR00
Number analyzed (Participants) | 77 | 73 | 79
Percent
  Cystoid Macular Edema | 0.0 | 0.0 | 1.3
  Hypopyon | 0.0 | 0.0 | 0.0
  Endolphthalmitis | 0.0 | 0.0 | 0.0
  Lens dislocated from posterior chamber | 0.0 | 0.0 | 0.0
  Pupillary block | 0.0 | 0.0 | 0.0
  Retinal detachment | 0.0 | 1.4 | 0.0
  Eyes with secondary surgical intervention | 1.3 | 4.1 | 1.3
Statistical Analysis 1: Comparison: Tecnis ZQR00; Test type: Superiority — Compare if study AE rate is significantly higher than ISO SPE rate (0.3% for retinal detachment); p = 0.1969, Exact test on binomial distribution — For ZQR00 retinal detachment
Statistical Analysis 2: Comparison: Tecnis ZHR00; Test type: Superiority — Compare if study AE rate is significantly higher than ISO SPE rate (0.8% for secondary surgical intervention); p = 0.4655, Exact test of binomial distribution — For ZHR00 secondary surgical intervention
Statistical Analysis 3: Comparison: Tecnis ZQR00; Test type: Superiority — Compare if study AE rate is significantly higher than ISO SPE rate (0.8% for secondary surgical intervention); p = 0.0210, Exact test on binomial distribution — For ZQR00 secondary surgical intention
Statistical Analysis 4: Comparison: Tecnis ZXR00; Test type: Superiority — Compare if study AE rate is significantly higher than ISO SPE rate (0.8% for secondary surgical intervention); p = 0.4698, Exact test on binomial distribution — For ZXR00 secondary surgical intervention

ADVERSE EVENTS:
Time Frame: 6 months
Description: The frequency and proportion of first eyes, second eyes and all subjects with these events is reported by IOL group.
  One subject had ZQR00 implanted in first eye and ZHR00 in second eye. For AE table this subject is included in both the ZQR00 and ZHR00 population group.
Groups:
- ZQR00: Investigational Lens Device
- ZXR00: Control Lens Device
Arm/Group | Tecnis ZHR00 | ZQR00 | ZXR00
All-Cause Mortality (participants affected / at risk) | 2/78 | 0/73 | 1/79
Serious Adverse Events (participants affected / at risk) | 8/78 | 7/73 | 5/79
Other Adverse Events (participants affected / at risk) | 4/78 | 3/73 | 3/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecnis ZHR00 (N=78) | ZQR00 (N=73) | ZXR00 (N=79)
Retinal tear and repair (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Clot in leg requiring emergency angioplasty (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary Surgical Intervention: IOL removal (Product Issues) | 1 (1) | 1 (2) | 1 (2)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia Surgical repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis of Large intestine with perforation resulting in hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lens removal due to undesired optical phenomena due to fixed pupil (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Heart Attack (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Death during sleep (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to surgical removal of tumors (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Death secondary to cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hospitalization due to weakness secondary to cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hospitalization due to hip fracture secondary to fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecnis ZHR00 (N=78) | ZQR00 (N=73) | ZXR00 (N=79)
ADE, Bothersome visual symptoms causing significant impairment lasting more than 3 mos postop (Product Issues) | 4 (4) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03111550/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03111550/SAP_001.pdf